CLINICAL TRIAL: NCT06406777
Title: Validation of MRI, CT and Pulmonary Function Tests for Early Detection of Chronic Lung Allograft Dysfunction
Brief Title: Chronic Lung Allograft Dysfunction MRI Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sean Fain (Other)
Responsible Party: Sponsor-Investigator, Sean Fain, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202304226
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Chronic Lung Allograft Dysfunction Lung MRI (CLAD)
Keywords: Lung Transplant
MeSH Terms: interventions — Spirometry; Radionuclide Imaging

STUDY DESIGN:
Intervention Model Description: Three populations that will all have the same interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Normal Subjects (Active Comparator): Healthy subjects, with no lung diagnosis, who are non-smokers.
  Interventions: Diagnostic Test: Spirometry; Diagnostic Test: Contrast Lung Computed Tomography (CT) Scan; Diagnostic Test: Oxygen enhanced magnetic resonance imaging (OE-MRI) Scan; Drug: 129Xe MRI scans
- Post Lung Transplant with normal functioning (Experimental): Subjects who have had a lung transplant and now have normal lung function
  Interventions: Diagnostic Test: Spirometry; Diagnostic Test: Contrast Lung Computed Tomography (CT) Scan; Diagnostic Test: Oxygen enhanced magnetic resonance imaging (OE-MRI) Scan; Drug: 129Xe MRI scans
- Post Lung Transplant with Chronic Lung Allograft Dysfunction (CLAD) (Experimental): Subjects who have had a lung transplant that now have CLAD
  Interventions: Diagnostic Test: Spirometry; Diagnostic Test: Contrast Lung Computed Tomography (CT) Scan; Diagnostic Test: Oxygen enhanced magnetic resonance imaging (OE-MRI) Scan; Drug: 129Xe MRI scans

INTERVENTIONS:
Diagnostic Test: Spirometry — Spirometry measures lung function, specifically the amount and/or speed of air that can be inhaled and exhaled.
Diagnostic Test: Contrast Lung Computed Tomography (CT) Scan — CT scan of the lungs using contrast
Diagnostic Test: Oxygen enhanced magnetic resonance imaging (OE-MRI) Scan — MRI will be taken while subject is lying on their back breathing 100% oxygen.
Drug: 129Xe MRI scans — MRI will be taken while subject is lying on their back breathing room oxygen and taking a breath of 129Xe and holding it for a few seconds.

SUMMARY:
This studies purpose is to confirm the efficacy and efficiency of using OE-MRI and MRI with hyperpolarized gas techniques and Iodinated contrast CT scan, this will enhance understanding of CLAD pathophysiology. Moreover, this project is foundational to performing additional studies to establish if novel MRI imaging can serve as an objective confirmatory diagnostic tool for CLAD in post-transplant patients.

DETAILED DESCRIPTION:
This studies purpose is to confirm the efficacy and efficiency of using OE-MRI and MRI with hyperpolarized gas techniques and Iodinated contrast CT scan, this will enhance understanding of CLAD pathophysiology. Moreover, this project is foundational to performing additional studies to establish if novel MRI imaging can serve as an objective confirmatory diagnostic tool for CLAD in post-transplant patients.

This observational imaging study will use 3T UTE MRI with varying oxygen levels (room air vs. 100% oxygen) to evaluate lung ventilation using oxygen enhanced imaging, in 50 healthy normal subjects (age 18-80).

Subjects will have vital signs taken, complete questionnaires and have pulmonary function test (spirometry) done, Iodinated contrast CT scan and standard of care CT scans, in addition to one MRI session that will include 6 series of scans. The MRI scans will be taken in supine position (laying on back) and include breathing room air and 100% oxygen. OE-MRI will be done in addition to MRI scans with Xenon-129.

ELIGIBILITY:
All subjects-Inclusion Criteria:

* Ages 18-80
* English Speaking Subjects
* Willingness and ability to provide informed consent
* Non-smoker

Lung transplant patients-inclusion criteria:

* >/= 6 months from lung transplant
* History of bilateral lung transplant

CLAD-free patients-inclusion criteria:

* Stable spirometry with FEV1 > 90% of baseline value (average of 2 best values) and forced mid-expiratory flow (FEF) (25-75) > 75% of baseline
* Total Lung Capacity (TLC) > 90 % of baseline
* Post-transplant chest radiograph without significant abnormality
* No evidence of on-going lung infection or allograft rejection

Early CLAD patients-inclusion criteria:

* FEV1 < 80% of baseline value (average of 2 best values)
* Follow up 6-months or decline in lung function (20% decrease in FEV1 without evidence of infection or acute rejection)

Exclusion Criteria:

* SAO2 drops below 90% (in absence of mechanical failure) during normal tidal breathing
* Unilateral diaphragm paralysis
* Evidence of acute illness on day of study
* Evidence of restrictive lung disease
* Dependence on supplemental oxygen
* History of cardiac disease
* Pregnancy (self-declared)
* Lactating women
* Participants with metal objects in their body
* Known contraindication to MRI examination
* Systolic blood pressure reading of < 100 mmHg or > 200 mmHg
* Diastolic blood pressure reading of <60 mmHg or > 100 mmHg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) Decline | Baseline and 3 months
  Absolute decrease of FEV1 by 20%

CONTACTS AND LOCATIONS:
Overall Officials: Sean Fain, Ph.D, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States